CLINICAL TRIAL: NCT04885465
Title: Web-based Support to Caregivers Supporting a Person With Heart Failure - a Randomised Controlled Trial With a Process Evaluation
Brief Title: Web-based Support to Caregivers in Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anna Stroemberg, professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Dnr 2019-05310
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Family Caregivers
Keywords: heart failure; caregiver; carer; preparedness; Perceived control
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Study participants will receive a web-based support program
  Interventions: Behavioral: web-based psychoeducational support
- Control group waiting list (No Intervention): Study participants in the control group waiting list will receive standard support from health care and municipalities. After study termination they will receive access to the same web-based program as the experimental group

INTERVENTIONS:
Behavioral: web-based psychoeducational support — Caregivers in the experimental group will have access to psycho-educational support through a web-based plattform during 3 months.
  Arms: Intervention group

SUMMARY:
Caregivers of people with heart failure experience a lack of support from health care in their caring role. They often want to become more involved in care, receive education and have the opportunity to share experiences with other caregivers.

Objectives and hypothesis: Our hypothesis is that an internet-based support program that is developed in collaboration with caregivers of people with heart failure will increase preparedness to care (Preparedness for Caregiving Scale). We will also evaluate the effects of the support program on the experiences of caring including positive experiences and the impact of care on health and lifestyle (Caregiver Competence Scale, Rewards of Caregiving Scale, Heart Failure-Caregiver Questionnaire) and their management of heart failure (knowledge of heart failure, support for heart failure self-care and perceived control over heart disease). We will also explore if the patients' healthcare consumption is altered when caregivers receive more support.

Method: The project is a randomized controlled study where 300 caregivers from four health care regions will be randomised to either receive a support program via 1177 care guide or to a control group waiting list who receive standard support from health care and municipalities. After the termination of the study participants in the control group will also be offered access to the support program. Data will be collected with questionnaires at baseline and after 3 and 6 months. A process evaluation with semi-structured interviews to describe the relatives' experiences of using the program with be conducted.

Relevance: Caregivers have been involved in all stages of the development of the Internet-based support program. The evaluation focuses on both the effects of the intervention and factors that affect implementation and equality. Caregiver support that is delivered through 1177 care guide enables a more equal, efficient and accessible support for caregivers.

ELIGIBILITY:
Inclusion Criteria:

* A close relative identified by the patient who cares for, supports or helps this patient with a verified heart failure diagnosis ICD codes within I42 or I50 (i.e. all types of heart failure).

Exclusion Criteria:

* Relatives who are unable to carry out the data collection or participate in intervention (e.g. non-Swedish speaking, cognitive problems, severe mental illness, addiction)
* The patient or the close relative have a serious disease with expected short survival of < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 3 months in preparedness to care for a person with heart failure | Measured at baseline, after 3 months
  Total score of the Preparedness for Caregiving Scale including 8 items, min score 0, max score 32, higher score indicate better preparedness

SECONDARY OUTCOMES:
Change from baseline to 3 and 6 months in Rewards of Caregiving | Measured at baseline, after 3 and 6 months
  Total score of the Rewards of Caregiving Scale including 10 items, min score 0, max score 40, higher score indicate better Rewards of caregiving
Change from baseline to 3 and 6 months in Caregiver Competence | Measured at baseline, after 3 and 6 months
  Total score of the Caregiver Competence Scale, including 4 item, min score 0, max score 12, higher score indicate better Caregiver Competence
Heart Failure-Caregiver burden and stress | Measured at baseline, after 3 and 6 months
  Total score and subscales of the Heart Failure-Caregiver Questionnaire including 21 item in three domains, namely physical (five items), emotional/psychological (11 items) and lifestyle (four items and one stem item). Items are scored on a severity response scale ranging from 'Not at all = 0' to 'A lot = 4'. The total score was the average of the sum of the three domain scores calculated from sum of scores for items answered/total possible score of items answered x 100. The minimum and maximum scores ranged between 0 and 100.Higher score indicate higher caregiver burden.
Perceived control over the heart disease | Measured at baseline, after 3 and 6 months
  Total score of the Control Attitude scale- caregiver version 4 item, min score 4, max score 28, higher score indicate better perceived control
Change from baseline to 6 months in preparedness to care for a person with heart failure | Measured at baseline, after 6 months
  Total score of the the Preparedness for Caregiving Scale including 8 items, min score 0, max score 32, higher score indicate better preparedness
Change in knowledge about heart failure in the three subscales | Measured after 3 months
  Revised Dutch heart failure knowledge scale with 3 subscales: 1. Knowledge subscale 15 items, min score 0 max score 15, higher score indicate better heart failure knowledge. 2. Trust in own HF knowledge subscale 3 items, min score 3 max score 15, higher score indicare better trust. 3. Health literacy subscale 3 items, min score 3 max score 15, higher score indicare better health literacy.
Change in caregiver support for heart failure self-care | Measured at baseline, after 3 and 6 months
  European Self-care Behaviour Scale - caregiverversion 7 items, Score from 0-100, higher score better support for self-care

OTHER OUTCOMES:
Social support | Measured at baseline, after 3 and 6 months
  Multidimensional Scale of Perceived Social Support, 12 items. Each item is rated on a seven-point Likert-type response format (1 = very strongly disagree; 7 = very strongly agree). A total score is calculated by summing the results for all items. The possible score range is between 12 and 84, the higher the score the higher the perceived social support.
Symptoms of anxiety and depression | Measured at baseline, after 3 and 6 months
  Hospital anxiety and depression scale, 7 items for anxiety and 7 items for depression. Min score 0 and max score 21 for each scale, Higher score indicate more symptoms of anxiety and depression
Health related quality of life | Measured at baseline, after 3 and 6 months
  EuroQol EQ-5D 5 level, index and VAS 0-100, higher score indicate better health

CONTACTS AND LOCATIONS:
Overall Officials: Anna Strömberg, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University Hospital, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No